CLINICAL TRIAL: NCT00180141
Title: Control of Therapy With Elidel vs Placebo in Patients With Atopic Dermatitis Using Bioengineering Methods
Brief Title: Elidel-Study: Elidel in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Roland Aschoff, MD, Technical University Dresden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981CDE16
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis on both lower arm.
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Elidel-Creme

SUMMARY:
Atopic dermatitis is a common disease. Emollients and Elidel have both shown to be effective to treat this disease. The research question is, whether the effective component (Elidel) is better than the emollient to improve the skin function.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Atopic dermatitis on both lower arms at least 1% body surface area.
* Atopic Dermatitis Severity Index (ADSI)-Score >= 6
* Investigator Global Assessment (IGA)-Score >= 2

Exclusion Criteria:

* Systemic therapy with immunosuppressive drugs within the past 24 weeks
* Phototherapy against atopic dermatitis.
* Antibiotic therapy against atopic dermatitis.
* Allergy against Elidel.
* Pregnancy
* Nursing
* Skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Aschoff, MD, Principal Investigator — Department of Dermatology. Medical Faculty, Technical University Dresden, Germany
Locations (1):
- Technical University Dresden, Dresden, Saxony, Germany